CLINICAL TRIAL: NCT05623904
Title: Carotid Revascularization Versus Best Medical Treatment for Asymptomatic Carotid Stenosis: a Multicenter, Open, Randomized Controlled Trial in Chinese Population
Brief Title: Carotid Revascularization Versus Best Medical Treatment for Asymptomatic Carotid Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: China-Japan Friendship Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Changhai Hospital (Other); Peking Union Medical College Hospital (Other); Hebei General Hospital (Other); The Second Hospital of Hebei Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Fifth Affiliated Hospital of Zhengzhou University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRBMACS
Record Dates: First submitted 2022-10-09; First posted 2022-11-21 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-12

CONDITIONS: Carotid Artery Stenting; Carotid Endarterectomy; Best Medical Treatment; Carotid Artery Stenosis Asymptomatic
Keywords: Carotid Revascularization; Carotid Artery Stenting; Carotid Endarterectomy; Best Medical Treatment; Carotid Artery Stenosis Asymptomatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carotid Revascularization (Active Comparator): Carotid Artery Stenting/Carotid endarterectomy + Best Medical Treatment
  Interventions: Procedure: Carotid Revascularization; Drug: Medical Treatment
- Medical Treatment (Active Comparator): Best Medical Treatment
  Interventions: Drug: Medical Treatment

INTERVENTIONS:
Procedure: Carotid Revascularization — Carotid Artery Stenting/Carotid Endarterectomy
  Arms: Carotid Revascularization
Drug: Medical Treatment — Aspirin 100mg/ day plus clopidogrel 75mg/ day for the first three months after enrollment or revascularization, aspirin 100mg/ day after three months, and the statin dose was adjusted according to blood lipids levels. Best medical treatment also includes risk factor control: good lifestyle, smoking cessation, weight control, regular exercise, SBP < 140 mmHg, HDL < 70 mg/dl (1.8mmol/L), and glycemic control. Patients with poor control of risk factors were dynamically adjusted during follow-up.
  In addition, patients undergoing CAS received dual antiplatelet therapy for at least 3 to 5 days before surgery, and patients undergoing CEA also received a preoperative oral antiplatelet drug (aspirin 100mg/ day, or clopidogrel 75mg/ day) for at least 3 days after enrollment.

SUMMARY:
This is a multicenter, open, randomized controlled trial to evaluate the efficacy and safety of carotid artery stenting/carotid endarterectomy versus best medical treatment for asymptomatic carotid artery stenosis in Chinese population.

DETAILED DESCRIPTION:
This is a multicenter, open, randomized controlled trial to evaluate the efficacy and safety of carotid artery stenting/carotid endarterectomy versus best medical treatment for asymptomatic carotid artery stenosis in Chinese population. The study will be conducted at 11 centers and is expected to enroll 1056 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years;
2. Carotid artery stenosis 50%-90% (ultrasound, CT, or DSA);
3. Asymptomatic carotid stenosis, that is, no transient ischemic attack, stroke, or other neurological symptoms in the past 6 months;
4. Patients who could complete 12 months of follow-up;
5. Patients who signed informed consent forms.

Exclusion Criteria:

1. Patients who had a TIA, stroke, or other related neurological symptoms within the previous 6 months;
2. Patients with spontaneous intracerebral hemorrhage in the past 12 months；
3. Patients with large intracranial aneurysms (diameter> 5mm)，and cannot be treated in advance or contemporaneous;
4. Chronic total occlusion without obvious cerebral ischemia symptoms；
5. Patients with neurologic disorder that caused transient or permanent neurological deficits and can not be identified with transient ischemic attack or stroke；
6. Patients with severe dementia;
7. Common carotid artery opening lesion；
8. Severe intracranial stenosis in tandem;
9. Carotid artery dissection;
10. Carotid artery aneurysm;
11. Myocardial infarction occurred within 30 days；
12. It is known that two or more proximal or main coronary artery stenosis ≥70%, untreated or unable to recanalize;
13. Ejection fraction <30% or New York Heart Association (NYHA) functional class III or higher；Unstable angina，ie angina at resting state and electrocardiogram changes；
14. Patients with cardiac emboli sources, such as left ventricular aneurysm, intraluminal filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, infective endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma；
15. Platelet count <5×104/μL, INR>1.5, Bleeding time > 1 min, or heparin-related thrombocytopenia；Patients contraindicated to heparin and antiplatelet drugs;
16. Patients with coagulation dysfunction.
17. Poor control of diabetes, fasting blood glucose >22mmol/L and ketone body > +2；
18. Malignant tumor or respiratory insufficiency, life expectancy < 5 years.
19. Insufficiency of vital organs: forced expiratory volume at one second < 30% (predicted)； dialysis-dependent renal failure; intolerance to anesthesia;
20. Currently waiting main organ transplants (ie heart, lung, liver, kidney), or are doing relevant evaluate；
21. Need to perform other general anesthesia surgery during the same period；
22. Pregnant or lactating women；
23. Those who participated in clinical trials of other drugs or medical devices before the inclusion did not reach the end of the time limit；
24. Investigators consider the patient inappropriate to participate in this clinical trial；

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Any Periprocedural Stroke, Myocardial Infarction, or Death During1 month Peri-procedural Period, and Postprocedural Ipsilateral Stroke 1 to 12-months. | 0 to 12 months
  Composite of any periprocedural stroke (ipsilateral or contralateral; major or minor), myocardial infarction, or death during1 month peri-procedural period, and postprocedural ipsilateral stroke 1 to 12-months.

SECONDARY OUTCOMES:
Technical success rate | 1 day
  Technical success was defined as final residual stenosis less than 30%, TIMI grade 3, and no dissection or thrombus after any endovascular treatment.
Rate of complications | 30 days
  Rate of complications within 30 days, complications include：Cranial nerve and peripheral nerve injury, vascular injury, non cerebral hemorrhage, wound complications as neck incision or related to puncture site, and other (such as anesthesia) complications.
Incidence of myocardial infarction | 30 days
  Incidence of myocardial infarction at 30 days follow up.
Incidence of ipsilateral stroke | 30 days
  Incidence of ipsilateral stroke at 30 days follow up.
Incidence of death | 30 days
  Incidence of death at 30 days follow up.
Carotid restenosis rate | 12 months
  Carotid restenosis was defined as restenosis ≥50% after carotid revascularization, that is, peak systolic velocity ratio (PSVR) ≥2.0 on ultrasound examination.
Incidence of target lesion revascularization | 12 months
  Target lesion revascularization (TLR) is defined as the re-percutaneous intervention or bypass grafting of the target lesion for restenosis or other complications of the target lesion. All TLR should be preclassified as clinically drived or non-clinically drived before the investigator performs angiography again.
Improvement in cognitive function | 30 days
  Cognitive function was assessed by Montreal Cognitive Assessment Scale (MoCA) at 30 days follow up.
Improvement in cognitive function | 30 days
  Cognitive function was assessed by Mini-mental State Examination (MMSE) at 30 days follow up.
Improvement in cognitive function | 12 months
  Cognitive function was assessed by Montreal Cognitive Assessment Scale (MoCA) at 12 months follow up.
Improvement in cognitive function | 12 months
  Cognitive function was assessed by Mini-mental State Examination (MMSE) at 12 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Gu, Dr., Principal Investigator — Xuanwu Hospital, Beijing
Locations (11):
- China (11):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided